CLINICAL TRIAL: NCT04981314
Title: Study on the Effect of an Echinacea Formulation on the Clinical Manifestations and Evolution of Covid-19
Brief Title: Echinacea Drug for Covid-19
Acronym: ECCO-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jesús R. Requena (Other)
Collaborators: IDIS (Unknown); SALUD (Unknown); Laboratoires Arkopharma (Industry)
Responsible Party: Sponsor-Investigator, Jesús R. Requena, Associate Professor, University of Santiago de Compostela
Organization: University of Santiago de Compostela (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-000850-24; 2021-000850-24 (EudraCT Number)
Record Dates: First submitted 2021-07-26; First posted 2021-07-29 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: Covid-19,; Echinacea
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Double blind, placebo controlled, randomised.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatments & placebos are coded. The code will not be revealed to investigators until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with echinacea (Experimental): EQUINÁCEA ARKOPHARMA, 2 caplets at breakfast, 2 caplets at lunch and 2 caplets at dinner with a glass of water, for 10 days.
  Interventions: Drug: Equinacea Arkopharma
- Placebo (Placebo Comparator): Hard caplets indistinguishable from EQUINÁCEA ARKOPHARMA, 2 caplets at breakfast, 2 caplets at lunch and 2 caplets at dinner with a glass of water, for 10 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Equinacea Arkopharma — Echinacea hard caplets
  Other Names: Echynacea hard caplets
  Arms: Treatment with echinacea
Other: Placebo — Placebo hard caplets
  Arms: Placebo

SUMMARY:
The main objectives of ECCO-2 are: 1) Efficacy: to study whether EQUINACEA ARKOPHARMA, hard caplets containing cryogenized root of the plant Echinacea purpurea, show an improvement of the clinical manifestations and disease course in ambulatory patients with covid-19 with a respiratory presentation and not requiring hospitalization (i.e., mild covid-19). The drug being evaluated will be added as a supplement of the standard treatment, with its current recommended dose for treatment of the common cold. 2) Safety: to determine that the incidence of adverse events is not higher than that seen with the standard treatment applied in each case.

DETAILED DESCRIPTION:
Different presentations of the plant Echinacea purpurea are widely prescribed and used for the treatment of upper respiratory tract viral infections. The plant is known to contain an array of active principles including alkylamides, cichoric acid, glucoproteins resulting in stimulation of the innate immune system, in particular, an activation of macrophages and an increase of phagocytic activity (Nagoor Meeran et al. 2019. Heliyon, 7(2):e05990). It has also been recently shown to exert a direct antiviral effect against SARS-CoV-II in vitro (Signer et al. 2020. Virol J 17:136). EQUINACEA ARKOPHARMA is a pharmaceutical preparation of Echinacea purpurea prepared by controlled cryo-processing roots of the plant and packing the powder thus obtained in hard caplets. The product is a medicine approved by the European Medicines Agency for the treatment of common cold. In this study, 230 patients presenting with mild Covid-19 at the emergency room of 4 participating hospitals, with an eminently respiratory presentation, fever, and not requiring hospitalization, will be randomly assigned to two branches to receive EQUINACEA ARKOPHARMA or placebo, in a double-blind manner. Patients will be followed up for 4 weeks and the effect of treatment vs. placebo on clinical manifestations, duration of fever and of total disease and percentage of return to the emergency room and/or hospitalization will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 99 años, with capacity to provide informed consent.
* Covid-19 diagnose, confirmed by PCR or antigen test
* Predominantly respiratory presentation. Additional minor digestive or/and neurological clinical manifestations will not lead to exclusion.
* Axillary temperature equal to or higher than 37ºC, at some point during the evolution of clinical signs prior to recruitment, or at the moment of recruitment.
* Being between days 1 and 9 of evolution of the disease, counting from the inception of symptoms.
* Not having received any Covid-19 vaccine.
* Capacity to complete the treatment, i.e., not having any swallowing difficulties, or any physical or psychiatric condition that would prevent the patient from taking caplets.
* Patients that after being evaluated at the emergency room are deemed to be in a condition to follow treatment at home, with follow up by their family doctor, i.e., that will not be hospitalized.

Exclusion Criteria:

* Patients under 18.
* Patients without a PCR or antigen test-based diagnose.
* Asymptomatic patients.
* Patients with an evolution higher than 9 days after the inception of symptoms
* Patients with a predominantly digestive presentation.
* Patients with a hypersensitivity to the active principle, any of the excipients of the drug or to the Asteraceae family of plants.
* Patients with systemic progressive diseases such as tuberculosis, diseases of the immune system, collagenosis, multiple sclerosis múltiple, AIDS, VIH infections and other immune diseases
* Patients previously treated at home with oxygen therapy.
* Non-collaborating patients.
* Patients without capacity to provide informed consent.
* Pregnant or nursing patients.
* Patients with an active immunosupressive treatment.
* Women in a potentially fertile age will need to provide a negative pregnancy test before being including in the study. Subsequently, they will be instructed about the convenience of not becoming pregnant during the study. Only women using reliable birth control measures will be included. WOCBPs unable to guarantee reliable birth control during the study, or using unreliable methods such as coitus interruptus, nursing or just spermicides, will be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Fever | 4 weeks since recruitment
  Number of days with fever equal or higher to 37 C

SECONDARY OUTCOMES:
Dyspnea | 4 weeks since recruitment
  Number of days with subjective dyspnea
Desaturation | 4 weeks since recruitment
  Number of days with desaturation (equal or less than 96%, measured with pulseoximeter provided)
Disease duration | 4 weeks since recruitment
  Days of disease duration
Hospitalizations | 4 weeks since recruitment
  Percentage of hospitalizations
Time of hospitalization | 4 weeks since recruitment
  Number of hospitalization days
Home sick leave days | 4 weeks since recruitment
  Number of home sick leave days
Emergency room visits | 4 weeks since recruitment
  Number of additional emergency room visits
Intensive Care Unit incoming | 4 weeks since recruitment
  Percentage of incoming to ICU
Deaths | 4 weeks since recruitment
  Percentage of deaths
Recruiter´s subjective improvement impression | 4 weeks since recruitment
  Score of recruiter´s subjective improvement impression
Patient´s subjective improvement impression | 4 weeks since recruitment
  Score of patient´s subjective improvement impression
Adverse events | 4 weeks since recruitment
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Pérez-Albiac, Study Chair — SALUD (Servicio Aragonés de Salud), Spain
Locations (4):
- Spain (4):
  - Hospital de Barbastro, Barbastro
  - Hospital do Barbanza, Ribeira
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Main results will be submitted for publication in a biomedical journal. The remaining IPD will be made availble to researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One month after study completion.
Access Criteria: Biomedical community.